CLINICAL TRIAL: NCT04579809
Title: Results of Flexor Tendon Repair of the Hand in Children Below Six Yera Sof Age
Brief Title: Results of Flexor Tendon Repair of the Hand in Children Below Six Years of Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Hossny fawzy nakhla, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Flexor tendon repair in child
Record Dates: First submitted 2020-09-24; First posted 2020-10-08 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Flexor Tendon Rupture

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- children below six years (Active Comparator): children below sex years both genders
  Interventions: Procedure: 4 strand technique
- cooperative children (Active Comparator): repair of the tendos by modified kessler
  Interventions: Procedure: 4 strand technique

INTERVENTIONS:
Procedure: 4 strand technique — 4 strand technique reapir of tendin flexor injury

SUMMARY:
The incidence of flexor tendon injuries in pediatric patients has remained largely undocumented, with a frequency of 3.6 per 100 000 persons per year.The pediatric literature demonstrates a higher prevalence of flexor tendon injuries in men, caused by sharp objects (glass or knife)

DETAILED DESCRIPTION:
The diagnosis of flexor tendon injuries is more challenging in younger children than in adults . and delayed diagnosis in children is common . An innocuous appearing skin wound and a subtle functional deficit may hinder both presentation and identification of the injury.Pediatric flexor tendon injuries heal rapidly and contractures are rare, as long as the joint has not been injured. but Inadequate management can result in loss of hand function .

Data involving children rehabilitation remain unclear, with some studies showing no difference between early rehabilitation protocols and four weeks of cast immobilization . Some studies claim that protocols are not necessary in children younger than six years of age, and that only immobilization is required and some studies show transition to a more aggressive early motion protocol .

Although the incidince of flexor tendon injury in children is not low but the reported cases below the age of six years remains low Which makes reported results less trustworthy. This created the need for a better designed and larger number study to report results in this age group.

ELIGIBILITY:
Inclusion Criteria:

* Acute flexor tendon injuries of the hand in both genders. All flexor zones are included. Cooperative patients aged between 0-6 years.

Exclusion Criteria:

* Uncooperative patients such as psychologically disturbed patients , who will not be able to follow the strict of protocol
* Age more than six years old .
* Associated fractures close to the tendon injury.
* Vascular injury requiring revascularization

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-12-25 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
range of motion of flexor tendon after repair according total active motion criteria | follow up the patients up to one year
  above elbow cast fo four weeks

REFERENCES:
- [Background] Piper SL, Wheeler LC, Mills JK, Ezaki M, Oishi SN. Outcomes After Primary Repair and Staged Reconstruction of Zone I and II Flexor Tendon Injuries in Children. J Pediatr Orthop. 2019 May/Jun;39(5):263-267. doi: 10.1097/BPO.0000000000000912. PMID 30969257